CLINICAL TRIAL: NCT01152541
Title: Corneal Collagen Crosslinking for Progressive Keratoconus and Ectasia Using Riboflavin/Dextran and Hypotonic Riboflavin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cornea and Laser Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYPO-CXL-001
Record Dates: First submitted 2010-06-22; First posted 2010-06-29 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Keratoconus; Corneal Ectasia
Keywords: Keratoconus; Corneal Ectasia; Collagen Crosslinking; Riboflavin
MeSH Terms: conditions — Keratoconus | interventions — Riboflavin; Dextrans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypotonic Riboflavin (Active Comparator): Administration of hypotonic riboflavin every 2 minutes for the duration of UV exposure.
  Interventions: Drug: Hypotonic Riboflavin
- Riboflavin/dextran (Active Comparator): Administration of Riboflavin/dextran every 2 minutes for the duration of UV exposure.
  Interventions: Drug: Riboflavin/Dextran

INTERVENTIONS:
Drug: Riboflavin/Dextran — Administration of riboflavin/dextran every 2 minutes for the duration of UV exposure
  Other Names: Riboflavin in a dextran solution
  Arms: Riboflavin/dextran
Drug: Hypotonic Riboflavin — Administration of hypotonic riboflavin every 2 minutes for the duration of UV exposure.
  Other Names: Hypotonic (low salt) riboflavin solution without dextran
  Arms: Hypotonic Riboflavin

SUMMARY:
Corneal collagen crosslinking (CXL) has been proposed as an effective method of reducing progression of both keratoconus and corneal ectasia after surgery, as well as possibly decreasing the steepness of the cornea in these pathologies. During the CXL procedure, the central corneal thickness has been shown to significantly change. The investigator's believe that better maintenance of corneal thickness potentially could have benefits of better reproducibility of the crosslinking effect with improved predictability of results.

DETAILED DESCRIPTION:
The objective of this study is to investigate the difference between the two riboflavin preparations during UV (ultraviolet) administration. Both riboflavin preparations currently are in general use worldwide and in U.S. clinical trials of corneal collagen crosslinking. The first preparation contains riboflavin in a dextran solution, which may tend to dehydrate the cornea and keep it thinner. The second preparation contains riboflavin in a solution without dextran; in this case, the relative hypotonicity may tend to keep the cornea better hydrated and thicker. The primary goal of the study is to see if the use of hypotonic riboflavin (rather than riboflavin with dextran) better maintains consistent corneal thickness during the CXL procedure. The second goal of the study is to determine if better maintenance of corneal thickness potentially could have benefits of better consistency of the procedure, decrease in corneal haze formation, and improved safety of the endothelial cells. Safety and efficacy outcomes will then be compared between the groups. In particular, we will compare the corneal thickness measured by ultrasonic pachymetry immediately after the CXL procedure in the randomized eyes. Secondary outcomes will include visual acuity, longer term corneal thickness changes, and corneal steepness changes. Safety assessments will include a tabulation of adverse events, patient symptoms, loss of visual acuity, changes in endothelial cell density, slit lamp examination of the cornea and lens, and contact lens tolerance for contact lens wearers

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* A diagnosis of progressive keratoconus over a period of 24 months or less before randomization or a diagnosis of corneal ectasia after corneal refractive surgery
* Vision with contact lenses or glasses is worse than 20/20
* Corneal thickness greater than 300 microns at the thinnest point

Exclusion Criteria:

* Eyes classified as either normal, atypical normal, or keratoconus suspect on the severity grading scheme.
* Corneal pachymetry ≤ 300 microns at the thinnest point measured by Pentacam in the eye(s) to be treated.
* Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications
* Clinically significant corneal scarring in the CXL treatment zone
* Pregnancy (including plan to become pregnant) or lactation during the course of the study
* A known sensitivity to study medications
* Patients with nystagmus or any other condition that would prevent a steady gaze during the CXL treatment or other diagnostic tests.
* Patients with a current condition that, in the investigator's opinion, would interfere with or prolong epithelial healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-06; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Corneal thickness | Intraoperatively
  Changes in central pachymetry (as measured by ultrasound) measured intraoperatively will be compared to a baseline preoperative value. Thickness will also be assessed at 1, 3, 6 and 12 months postoperatively.

SECONDARY OUTCOMES:
Maximum Keratometry | 12 months
  The change in maximum keratometry (Kmax) from baseline will be evaluated at 12 months for all eyes randomized to (Group 1 - administration of Riboflavin/dextran for the duration of UV exposure.) and (Group 2 - Administration of hypotonic riboflavin for the duration of UV exposure) groups. As a secondary analysis of this endpoint, the change in maximum keratometry (Kmax) from baseline will be evaluated at 1, 3 and 6 month for all eyes
Manifest Refraction | 12 months
  The change in manifest refraction spherical equivalent from baseline will be evaluated at 12 months. As a secondary analysis of this endpoint, a repeated measures analysis of variance will be conducted to assess the profile of the treatments across time at 1 month for the treatment groups as well as at 3, and 6 months to look at the effect of CXL timing on this variable.
Visual Acuity | 12 months
  Change in BSCVA (best spectacle corrected visual acuity) and UCVA (uncorrected visual acuity) compared to the baseline examination will be evaluated at 12 months postoperatively. As a secondary analysis of this endpoint will be conducted to assess the profile of the treatments across time at 1 month and again at 3, and 6 months following the CXL procedure.
Endothelial Cell Density | 12 months
  Endothelial cell count will be obtained using specular microscopy (Konan Medical) prior to CXL treatment and at 12 months postoperatively. Measurements will also be taken 3 months postoperatively and compared to baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hersh, MD, Principal Investigator — Cornea and Laser Eye Institute
Locations (1):
- Cornea and Laser Eye Institute, Teaneck, New Jersey, United States